CLINICAL TRIAL: NCT05847517
Title: Randomised, Double-blind, Placebo-controlled Clinical Trial to Evaluate the to Assess the Efficacy of Intravenous Metoprolol in Patients With Acute Respiratory Distress Syndrome (ARDS).
Brief Title: Metoprolol in Acute Respiratory Distress Syndrome (MAIDEN)
Acronym: MAIDEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: European Commission (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAIDEN
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: metoprolol; beta-blockers; sepsis; orotracheal intubation; Pathologic Processes; Respiratory Disease; Neutrophil Extracellular Traps; platelet aggregation; diffuse alveolar damage; neutrophil infiltration; Pulmonary Inflammation; pancreatitis; Severe Acute Respiratory Syndrome-Corona Virus-2; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis; Pathologic Processes; Respiration Disorders; Pneumonia; Pancreatitis; Drug-Related Side Effects and Adverse Reactions | interventions — Metoprolol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomization (1:1) will be stratified according to the severity of ARDS and by participating centre:
  * Moderate (PaO2/FiO2 of 100-200 mmHg).
  * Severe (PaO2/FiO2 ≤100 mmHg).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both metoprolol and saline are supplied in 5 ml ampoules of the same shape, structure and colour
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoprolol (Active Comparator): Participants will be administered IV Metoprolol tartrate 15 mg (3 ampoules of 5 ml) diluted in 100 ml of saline.
  Interventions: Drug: Metoprolol Injection
- Saline (Placebo Comparator): Participants will be administered IV saline (0.9% sodium chloride) (3 ampoules of 5 ml) diluted in 100 ml of saline.
  Interventions: Drug: saline 0.9%

INTERVENTIONS:
Drug: Metoprolol Injection — A dilution of 15 mg Metoprolol tartrate in 100 ml saline shall be performed and infused for 10 minutes. No dose reduction or increase is allowed. Systolic blood pressure and heart rate shall be measured 3 and 6 minutes after starting the infusion.
  In case of a consistent drop in systolic blood pressure or heart rate, the infusion shall be stopped and the infusion noted.
  Arms: Metoprolol
Drug: saline 0.9% — A dilution of 0.9% sodium chloride in 100 ml saline shall be performed and infused for 10 minutes. No dose reduction or increase is allowed. Systolic blood pressure and heart rate shall be measured 3 and 6 minutes after starting the infusion.
  In case of a consistent drop in systolic blood pressure below 110 mmHg or heart rate below 60 bpm, the infusion shall be stopped and the infusion noted.
  Arms: Saline

SUMMARY:
Randomised, double-blind, placebo-controlled clinical trial to evaluate the efficacy of intravenous metoprolol in patients with Acute Respiratory Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
This is a placebo-controlled, randomised, double-blind, multicentre, Phase III clinical trial to assess the efficacy of IV metoprolol in newly intubated ARDS patients, assessing survival and days free of invasive mechanical ventilation during the first 28 days. Eligible participants shall have had orotracheal intubation (OTI) and mechanical ventilation within 72 hours prior to randomisation, moderate-severe ARDS (PaO2/FiO2: ≤200 mmHg under standardised conditions (PEEP≥5 cm H2O), a heart rate ≥ 60 bpm and invasive systolic blood pressure ≥ 110 mmHg.The trial will include a total of n=350 patients, with two treatment arms: metoprolol vs. placebo (1:1). Each of the 7 days of treatment, participants will be receive 15 mg of iv metoprolol tartrate or matching placebo in 100 ml of saline for 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years and <80 years) with a clinical diagnosis of ARDS of any aetiology (pneumonia, including SARS-CoV-2, sepsis, pancreatitis, bronchospasm and trauma) admitted to the ICU.
* Orotracheal intubation (OTI) and mechanical ventilation within 72 hours prior to randomisation.
* Moderate-severe ARDS (PaO2/FiO2: ≤200 mmHg under standardised conditions (PEEP≥5 cm H2O).
* Heart rate ≥ 60 bpm.
* Invasive systolic blood pressure ≥ 110 mmHg.

Exclusion Criteria:

* Prolonged hospital admission prior to randomisation (i.e. ≥7 days at the time of randomisation).
* Reduced left ventricular ejection fraction (LVEF <50%).
* Life expectancy due to other processes (cancer, degenerative diseases, etc.) of less than 6 months.
* Right ventricular (RV) systolic dysfunction.
* Concomitant acute heart failure (cardiac index ≤2.5 L/m2 or pulmonary capillary pressure ≥15 mmHg or clinical suspicion).
* Second-degree atrioventricular (AV) block, 2:1 AV block, high-grade/advanced AV block and third-degree AV block. Also significant sinus bradycardia, which would be implied by having a heart rate >60 bpm as an inclusion criterion.
* Pregnant or breastfeeding women.
* Cardiogenic shock.
* Persistent invasive blood pressure <110 mmHg despite vasopressor agents.
* Use of noradrenaline at concentrations greater than 0.2 µg/kg/min at the time of the randomisation.
* Use of dobutamine within 48 hours before randomisation.
* Concomitant pulmonary embolism.
* Known severe peripheral arterial disease.
* Known asthma before admission (with active bronchodilator therapy).
* Active beta-blocker treatment prior to admission (i.e. within 3 months prior to admission).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
days alive and free of invasive mechanical ventilation during the first 28 days. | 28 days
  Hierarchical composite outcome "Alive and ventilator-free days at 28 days" (win ratio approach)

SECONDARY OUTCOMES:
All-cause death at day 28 after randomization | 28 days
  cumulative incidence of death from any cause
Ventilator-free days at 28 days | 28 days
  number of days without mechanical ventilation during the firs 28 days
Intensive care unit days of admission | 3 months
  Number of days admitted at the intensive care unit
Quality of life score | at 3 months
  Mean quality of life score according to ''The Short Form 36 Health Survey Questionnaire'' (SF-36). The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Arterial oxygenation | on day 8
  Mean arterial oxygen saturation (PaO2/FiO2)
Change in arterial oxygenation | 8 days
  Mean difference in arterial oxygen saturation (PaO2/FiO2) between baseline and day 8

CONTACTS AND LOCATIONS:
Overall Officials: Borja Ibanez, MD PhD FESC, Principal Investigator — CNIC & Fundación Jiménez Díaz University Hospital
Locations (10):
- Spain (10):
  - Hospital Universitario de Jerez de La Frontera, Jerez de la Frontera, CADIZ
  - Hospital Universitario de Toledo, Toledo, Castille-La Mancha
  - Hospital Clinic, Barcelona, Catalonia
  - Hospital Parc Taulí, Barcelona, Catalonia
  - Fundación Jiménez Díaz University Hospital, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital de Getafe, Madrid, Madrid
  - Hospital General de Villalba, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Rey Juan Carlos, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No